CLINICAL TRIAL: NCT00594399
Title: Enhancing Fitness in Older Overweight Vets With Impaired Fasting Glucose
Brief Title: Enhancing Fitness in Older Pre-diabetic Veterans
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 06-252
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-08

CONDITIONS: Impaired Glucose Tolerance; Obesity; Diabetes
Keywords: Aging; Exercise; Impaired Glucose Tolerance; Obesity; Functional Status; Disability; Health Services Research; Randomized Controlled Trial; Diabetes; Adaptive Randomization Design
MeSH Terms: conditions — Glucose Intolerance; Obesity; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Physical Activity counseling (Experimental): Physical activity (PA) counseling program with the following components: baseline in-person counseling session; telephone calls, one physician endorsement of PA in a primary care clinic visit, monthly automated telephone calls from the primary care provider encouraging PA; and quarterly mailed materials providing personalized feedback.
  Interventions: Behavioral: Physical Activity Counseling
- Arm 2 (No Intervention): Usual care from primary, womens or geriatric clinics

INTERVENTIONS:
Behavioral: Physical Activity Counseling — Physical activity (PA) counseling program with the following components: a baseline in-person counseling session; telephone calls biweekly for 6 weeks then monthly; one physician endorsement of PA in a primary care clinic visit; monthly automated telephone calls from the primary care provider encouraging PA; and (5) quarterly mailed materials providing personalized feedback.
  Arms: Arm 1 Physical Activity counseling

SUMMARY:
This study targets older adults (ages 60 and over) who are overweight (body mass index 25-40) with impaired fasting glucose (100 - 125). We propose a three-year, randomized controlled clinical trial (n=300) to determine the effect of a one-year physical activity counseling intervention on glucose metabolism and secondary outcomes compared to usual care.

DETAILED DESCRIPTION:
IMPACT. Our proposed project will contribute to improved quality and efficiency of VA health care by: (1) providing an effective program of Enhanced Fitness counseling that will result in a significant increase in physical activity of sufficient magnitude to achieve noted improvements in glycemic control, and (2) developing and disseminating materials that can be used throughout the VHA for physical activity promotion for older, overweight adults.

BACKGROUND. The nation is experiencing a marked increase in obesity, and diabetes. Users of the VA medical facilities report higher than national average rates of obesity and diabetes. Current projections indicate that 70% of veterans using the VA medical care are overweight, 20% have diabetes, and 30- 40 % have metabolic syndrome. Approximately 30 % of VA health care costs are attributable to care for diabetes alone. Incidence and prevalence of these conditions increase with age and are associated with high medical costs. This is especially true of the older adult who typically has added comorbidities and functional limitations. The VHA has aggressively addressed the existing epidemic by implementing various programs and performance measures aimed at attaining optimal medical management of dyslipidemia, diabetes, and obesity. The component of all of these initiatives that has received the least amount of attention is physical activity despite overwhelming evidence that physical activity can favorably alter all of the medical conditions described above. The VA system-wide has been ill equipped to provide feasible, cost effective physical activity programs despite the imperative to seek ways to reduce incident diabetes and reduce potential health care costs.

OBJECTIVES. We propose an innovative home-based enhanced fitness counseling intervention that involves a unique partnership between veteran, primary care provider, and exercise counselor directed at the older adult. The proposed project, Enhanced Fitness, seeks to improve glycemic control in older, overweight adults with impaired fasting glucose receiving primary care at the VA. A novel design, adaptive randomization, will allow us to assess the impact of our intervention at an early stage and then reassign individuals to a more intense or reduced intervention based upon patient compliance. Due to the national implementation of MOVE! in primary care for the treatment of obesity we will consider MOVE! as part of usual care for this population. Primary Hypothesis. Compared to usual care (plus MOVE!), individuals receiving Enhanced Fitness counseling will have significantly improved glucose metabolism (fasting insulin). Secondary Research Hypotheses and Objectives. (1) Compared to usual care (plus MOVE!), individuals receiving Enhanced Fitness counseling will have significantly improved secondary outcomes related glycemic control (fasting blood glucose, HOMA-IR, HbA1c, metabolic syndrome score), physical function (self report and physical performance), disability, and health related quality of life; and (2) To determine differences in cost and health care utilization between groups.

Note: 7/5/2010: An amendment was submitted and approved to drop the adaptive randomization component of the study. This was necessary due to low levels of noncompliance observed during the first follow-up assessment. The primary and secondary objectives of the study were not affected by this amendment.

Another amendment was submitted and approved to: 1) evaluate the association between APOE, diabetic risk and physical function; and 2) to examine associations between inflammatory markers, diabetic risk, and physical function.

METHODS: For the proposed study we will target older adults (ages 60 and over) who are overweight (body mass index >24-40) with impaired fasting glucose (100 - 125). We propose a three-year, randomized controlled clinical trial (n=300) to determine the effect of our 1-year Enhanced Fitness counseling intervention on glucose metabolism. A novel design, adaptive randomization, will allow us to mimic primary care by altering treatment based upon patient compliance. We will use a "train the trainers" approach for dissemination of results at the local, VISN, and national level.

ELIGIBILITY:
Inclusion Criteria:

* VA patients followed by the Durham VA Primary Care, Women's Health, and Geriatric clinics
* Must have had more than one visit to the VA in preceding 12 months
* Age 60 and over
* Impaired glucose intolerance documented by recent fasting blood glucose between 100 and 125 mg/dL
* Body mass index between 25-40 kg/m2
* Able to walk 10 meters without human assistance (assistive device acceptable)
* All participants must be assigned a primary care provider and have had more than one visit to the VA in the preceding 12 months

Exclusion Criteria:

* Free of frank diabetes
* Fasting blood sugar above 125 mg/dL
* HbA1c > 7%
* Unstable angina
* Recent history of ventricular tachycardia
* Unstable chronic obstructive pulmonary disease (two hospitalizations within the previous 12 months and/or on oxygen)
* Uncontrolled hypertension (diastolic blood pressure >110 mm/Hg or systolic > 200mm/Hg)
* Stroke with moderate to severe aphasia
* Diagnosis of chronic pain which may interfere with their ability to be physically active
* Diagnosis of unstable mental or behavioral disorder
* Diagnosis of memory loss or dementia
* Visual or hearing loss severe enough to interfere with ability to receive telephone counseling and review written materials
* Active substance abuse
* A terminal diagnosis
* Followed by VA for medications only
* Regularly, vigorously physically active for six months or longer.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam C. Morey, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Turer CB, Bernstein IH, Edelman DE, Yancy WS Jr. Low HDL predicts differential blood pressure effects from two weight-loss approaches: a secondary analysis of blood pressure from a randomized, clinical weight-loss trial. Diabetes Obes Metab. 2012 Apr;14(4):375-8. doi: 10.1111/j.1463-1326.2011.01531.x. Epub 2011 Dec 27. PMID 22059803
- [Result] Morey MC, Pieper CF, Edelman DE, Yancy WS Jr, Green JB, Lum H, Peterson MJ, Sloane R, Cowper PA, Bosworth HB, Huffman KM, Cavanaugh JT, Hall KS, Pearson MP, Taylor GA. Enhanced fitness: a randomized controlled trial of the effects of home-based physical activity counseling on glycemic control in older adults with prediabetes mellitus. J Am Geriatr Soc. 2012 Sep;60(9):1655-62. doi: 10.1111/j.1532-5415.2012.04119.x. PMID 22985140
- [Result] Hall KS, Pieper CF, Edelman DE, Yancy WS Jr, Green JB, Lum H, Peterson MJ, Sloane R, Cowper PA, Bosworth HB, Huffman KM, Cavanaugh JT, Chapman JG, Pearson MP, Howard TA, Ekelund CC, McCraw BL, Burrell JB, Taylor GA, Morey MC. Lessons learned when innovations go awry: a baseline description of a behavioral trial-the Enhancing Fitness in Older Overweight Veterans with Impaired Fasting Glucose study. Transl Behav Med. 2011 Nov;1(4):573-587. doi: 10.1007/s13142-011-0075-6. PMID 22866170
- [Result] Povsic TJ, Sloane R, Green JB, Zhou J, Pieper CF, Pearson MP, Peterson ED, Cohen HJ, Morey MC. Depletion of circulating progenitor cells precedes overt diabetes: a substudy from the VA enhanced fitness trial. J Diabetes Complications. 2013 Nov-Dec;27(6):633-6. doi: 10.1016/j.jdiacomp.2013.08.004. Epub 2013 Sep 19. PMID 24055327
- [Result] Hall KS, Beckham JC, Bosworth HB, Sloane R, Pieper CF, Morey MC. PTSD is negatively associated with physical performance and physical function in older overweight military Veterans. J Rehabil Res Dev. 2014;51(2):285-95. doi: 10.1682/JRRD.2013.04.0091. PMID 24933726
- [Result] Povsic TJ, Sloane R, Zhou J, Pieper CF, Pearson MP, Peterson ED, Green JB, Cohen HJ, Morey MC. Lower levels of circulating progenitor cells are associated with low physical function and performance in elderly men with impaired glucose tolerance: a pilot substudy from the VA Enhanced Fitness trial. J Gerontol A Biol Sci Med Sci. 2013 Dec;68(12):1559-66. doi: 10.1093/gerona/glt067. Epub 2013 May 16. PMID 23682163
- [Derived] Povsic TJ, Sloane R, Pieper CF, Pearson MP, Peterson ED, Cohen HJ, Morey MC. Endothelial Progenitor Cell Levels Predict Future Physical Function: An Exploratory Analysis From the VA Enhanced Fitness Study. J Gerontol A Biol Sci Med Sci. 2016 Mar;71(3):362-9. doi: 10.1093/gerona/glv180. Epub 2015 Oct 28. PMID 26511012

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2, Usual Care: Usual care from primary, womens or geriatric clinics
- Arm 3, Physical Activity Counseling, Reduced Dose: Upon rerandomization, individuals in this group continued to receive monthly physical activity counseling through 6 months which was then reduced to every other month during months 6-12.
Period: Initial 3 Month Counseling
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2, Usual Care | Arm 3, Physical Activity Counseling, Reduced Dose
Started | 180 | 122 | 0
Completed | 163 | 118 | 0
Not Completed | 17 | 4 | 0
Not completed — Not ready to exercise | 1 | 0 | 0
Not completed — Lack of Interest | 3 | 3 | 0
Not completed — Personal issues | 2 | 0 | 0
Not completed — Too busy | 7 | 1 | 0
Not completed — Pain | 2 | 0 | 0
Not completed — Moved | 1 | 0 | 0
Not completed — Family illness | 1 | 0 | 0
Period: Rerandomization Arm 1 Only
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2, Usual Care | Arm 3, Physical Activity Counseling, Reduced Dose
Started | 81 (Total sample in Arm 1 was rerandomized and allocated to remain in Arm 1 or assigned to Arm 3) | 118 | 82 (This sample reflects newly randomized study Arm)
Rerandomization | 81 (Rerandomized to continue to receive telephone calls every 2 weeks or at a reduced dose of 1/ month) | 114 | 82
Completed | 79 | 114 | 82
Not Completed | 2 | 4 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The average age of the sample was 67 year with a range of 60 to 89. Participant were in a normal usual walking speed for their ages but were at the 10th percentile in norms for six-minute walk distance indicating poor aerobic capacity for their age.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2 | Total
Number analyzed (Participants) | 180 | 122 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (6.3) | 67.7 (6.2) | 67.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 173 | 119 | 292
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 39 | 88
  White | 129 | 83 | 212
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
usual gait speed [Mean (Standard Deviation); unit: meters/second] — Normal walking speed over 4 meters
  meters/second | 1.24 (0.3) | 1.25 (0.3) | 1.24 (0.3)
Physical Function [Mean (Standard Deviation); unit: points] — Physical function was measured by self report using the physical function subscale of the SF-36. Scores range from 0 to 100 with a higher score indicating better functioning.
  points | 62.94 (20.97) | 63.97 (21.79) | 62.98 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Insulin
Description: Fasting Insulin analyzed at VA central laboratory by technicians not affiliated with study. Participants were instructed to refrain from eating or drinking anything except water and medications past midnight. A reminder call was placed the night before the scheduled appointment and fasting was verified by study personnel before appointed blood draws.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
uIU/ml | 10.26 (6.09) | 10.39 (8.58)

2. Primary Outcome: 3 Month Fasting Insulin
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
uIU/ml | 10.04 (7.21) | 10.45 (7.82)

3. Primary Outcome: 12 Month Fasting Insulin
Time Frame: 12 months
Population: All of the primary analyses reported here were based upon comparisons to physical activity counseling (Arm 1) versus usual care (Arm 2). No subgroup analyses within the intervention arm were conducted for this primary outcome report. The decision to analyze and report the data in Arm 1 in aggregate was done apriori during design of the study.
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
uIU/ml | 11.4 (6.84) | 10.28 (5.59)
Statistical Analysis 1: Comparison: Arm 1 Physical Activity Counseling vs Arm 2; Test type: Superiority or Other; p = 0.43, Mixed Models Analysis — Omnibus test of difference between groups over time with Bonferroni correction and adjustment for baseline value of insulin

4. Primary Outcome: Fasting Glucose
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
mg/dl | 110.51 (6.95) | 110.6 (7.1)

5. Primary Outcome: 3 Month Fasting Glucose
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
mg/dl | 106.96 (9.59) | 107.63 (9.62)

6. Primary Outcome: 12 Month Fasting Glucose
Time Frame: 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
mg/dl | 104.35 (9.62) | 104.38 (11.97)
Statistical Analysis 1: Comparison: Arm 1 Physical Activity Counseling vs Arm 2; Test type: Superiority or Other; p = 0.91, Mixed Models Analysis — Omnibus test of difference between groups over time with Bonferroni correction and adjustment for baseline value of glucose

7. Secondary Outcome: Physical Activity, Endurance
Description: Physical activity, endurance/aerobic activities by self-report from the CHAMPS questionnaire of physical activity for older adults.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
minutes per week | 73.39 (119.81) | 115.29 (183.66)

8. Secondary Outcome: Physical Activity, Endurance
Description: as for outcome 7
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
minutes per week | 124.3 (127.15) | 92.87 (115.01)

9. Secondary Outcome: Physical Activity, Endurance
Description: as for outcome 7
Time Frame: 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Number analyzed (Participants) | 180 | 122
minutes per week | 133.6 (136.47) | 112.62 (135.45)
Statistical Analysis 1: Comparison: Arm 1 Physical Activity Counseling vs Arm 2; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Omnibus test of difference between groups over time with adjustment for baseline value of physical activity

ADVERSE EVENTS:
Time Frame: At each wave of data collection
Arm/Group | Arm 1 Physical Activity Counseling | Arm 2
Serious Adverse Events (participants affected / at risk) | 26/180 | 11/122
Other Adverse Events (participants affected / at risk) | 158/180 | 50/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Physical Activity Counseling (N=180) | Arm 2 (N=122)
The patient experienced dizziness and radiating shoulder pain (Cardiac disorders) | 1 | 0
Pt was informed 2-3 months ago that he had a brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Saw PCP - had chest pain (Cardiac disorders) | 1 | 0
While blowing leaves in his yard, his feet got tangled & he fell (Injury, poisoning and procedural complications) | 0 | 1
Phlebitis (started 2 wks ago)--affected left leg (Musculoskeletal and connective tissue disorders) | 1 | 0
Admitted to the VA hospital for chest pain and SOB. (Cardiac disorders) | 1 | 0
Pt had left inguinal surgery (Surgical and medical procedures) | 1 | 0
Scheduled for a cath at his regional hospital. Kept as an inpatient due to bleeding. (Cardiac disorders) | 1 | 0
Developed a TIA The symptoms, (right sided numbness) (Nervous system disorders) | 1 | 0
Patient has a cough was admitted overnight because of flu virus. (Infections and infestations) | 1 | 0
When the RA checked CPRS for the patient's next schedule stated date of death (General disorders) | 0 | 1
One-third of patients left lung was removed. He was diagnosed with lung CA. (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Patient passed away from a recurrence of lung cancer. (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pt hospitalized for a recurrence of lung cancer. (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Patient had a PCP appt at the VA and presented with bradycardia/A-fib. . (Cardiac disorders) | 1 | 0
Pt was admitted for pharmacological treatment for paroxysmal A-fib. (Cardiac disorders) | 1 | 0
Husband was thrown to the wall behind him breaking his left femur. (Injury, poisoning and procedural complications) | 1 | 0
Pt had a planned surgery on his L carotid artery (Cardiac disorders) | 1 | 0
Patient had emergency gallbladder surgery (Surgical and medical procedures) | 1 | 0
He had "a lot of pain in his back and down his left leg." (Musculoskeletal and connective tissue disorders) | 1 | 0
Via CT scan at regular visit to pulmonologist, discovered blood clot in lung. out of breath. (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Complications of an elective surgery. (outside VA) (Injury, poisoning and procedural complications) | 1 | 0
Shortness of breath - diagnosed with a heart attack. (Cardiac disorders) | 0 | 1
Pt had a MVA. Abrasion on his forehead, neck pain, headache, nausea, and vomiting. (Injury, poisoning and procedural complications) | 1 | 0
Pt had been sick with a cough was hospitalized for Bronchitis (?) & SOB. (Infections and infestations) | 0 | 1
Inability to urinate brought pt to the ER. enlarged prostate (new) caused UTI (abx) (Renal and urinary disorders) | 0 | 1
Gallbladder surgery (Surgical and medical procedures) | 1 | 0
The patient was scheduled for a heart catherization. (Cardiac disorders) | 1 | 0
Patient had a cath due to unstable angina, followed by an angioplasty receiving four stents. . (Cardiac disorders) | 1 | 0
Pt experienced symptoms of heat stroke admitted for dehydration, palpitations (General disorders) | 1 | 0
Pt had a dizzy spell and fell. No injuries from fall but went to ED for follow-up. (Injury, poisoning and procedural complications) | 0 | 1
Patient had a staph infection in his right foot. (Infections and infestations) | 0 | 1
Got out of the bed and was walking towards the bathroom and fell out. (Injury, poisoning and procedural complications) | 0 | 1
Patient reported a serious gout episode. (Metabolism and nutrition disorders) | 0 | 1
Patient had outpatient surgery for bladder cancer (Surgical and medical procedures) | 1 | 0
Patient experienced a heart attack (Cardiac disorders) | 1 | 0
Patient had a C-spine fusion surgery. The next day the patient passed away. (Surgical and medical procedures) | 1 | 0
Pt had an elective AICD implant primarily for prevention (Cardiac disorders) | 1 | 0
Patient had left knee surgery . (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt was admitted to the VA for left knee infection. He had a left TKA done (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 Physical Activity Counseling (N=180) | Arm 2 (N=122)
Pt has been "hibernating" for 3 weeks- not feeling well and spending most time in bed (Psychiatric disorders) | 1 | 0
More pain in LB and knees the last weeks (Spinal stenosis, s/p surgery x 3, OA). (Musculoskeletal and connective tissue disorders) | 1 | 0
His LBP flared up when trying to change tires on his trailer. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had a UTI. (Renal and urinary disorders) | 1 | 0
Treated for prostatitis. (Infections and infestations) | 1 | 0
L ankle swelling with pain for about 3 weeks. Swelling has decreased Scheduled to see PCP next month (Musculoskeletal and connective tissue disorders) | 1 | 0
Weak a couple of days r/t the weather. "got real hot" laid off of some activities for a couple days (General disorders) | 1 | 0
Had the flu. Did not see an MD. Will play in a golf tournament today. (Infections and infestations) | 1 | 0
2-3 weeks ago was at commode. Got weak and fell over into basin. Bruise at naval. (Injury, poisoning and procedural complications) | 1 | 0
Hurt his back on the golf course. (Musculoskeletal and connective tissue disorders) | 1 | 0
Was cleaning out the garden, stepped on a brick and his leg slipped causing a fall. (Injury, poisoning and procedural complications) | 0 | 1
Walking on dune at beach, the sand shifted and he fell on left side and shoulder. (Injury, poisoning and procedural complications) | 0 | 1
Fell on the kitchen floor and hit knee due to the "intestinal flu" (Injury, poisoning and procedural complications) | 0 | 1
Was empting grass container and pulled a muscle in back. (Injury, poisoning and procedural complications) | 0 | 1
Fell and thrust right hand/little finger into door jamb, almost pulling finger off hand (Injury, poisoning and procedural complications) | 0 | 1
Sciatic nerve started acting up. (Congenital, familial and genetic disorders) | 0 | 1
Had surgery for reversal of ileostomy in Burlington, . The surgery went very well. (Surgical and medical procedures) | 1 | 0
Had an MRI done for left knee. Is waiting for a second opinion app. with ortho at the VA. (Musculoskeletal and connective tissue disorders) | 1 | 0
L knee started hurting and swelling after water aerobics yesterday. (Musculoskeletal and connective tissue disorders) | 1 | 0
Woke up w/ pain in L hip on Had it for 8 days, mostly in the morning (Musculoskeletal and connective tissue disorders) | 1 | 0
Injured the left knee during the water aerobic class (Injury, poisoning and procedural complications) | 1 | 0
Went VA ER for an URI - got antibiotics. (Renal and urinary disorders) | 1 | 0
Had a bad sinus infection. Fine now. (Infections and infestations) | 1 | 0
Pts. allergies flared up. (Immune system disorders) | 1 | 0
Had a cyst taken out on his forehead at the VA. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Has had a cold last 10 days. (Infections and infestations) | 1 | 0
Pt. has been dizzy/lightheaded, (comes/goes), for the last 2 weeks (General disorders) | 1 | 0
Temporarily lost feeling in right leg and fell on grass. This is nerve related and not new problem. (Nervous system disorders) | 1 | 0
Had laser surgery done on left leg on - planned procedure. Has had a nerve pain in left leg (Surgical and medical procedures) | 1 | 0
His lower back has been acting up the last two weeks. He has seen his "Back" MD and been in rehab (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt had outpatient carpal tunnel surgery on left hand at the VA. (Musculoskeletal and connective tissue disorders) | 1 | 0
About 5 months ago, had carpal tunnel repair surgery on left hand. (Surgical and medical procedures) | 1 | 0
Had to have an epidural "pain block" for his LB pain. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt. had an appt with ENT due to blood drainage from the right ear (Ear and labyrinth disorders) | 1 | 0
Has had the flu . Has not seen an MD. Feeling better but still coughing. (Infections and infestations) | 1 | 0
Has had the flu. Has not seen the MD. (Infections and infestations) | 1 | 0
Got a crick in my neck. (Musculoskeletal and connective tissue disorders) | 0 | 1
Presented to the VA ER for left sided chest pain/ arm/leg pain radicular from his spinal stenosis. (Musculoskeletal and connective tissue disorders) | 1 | 0
Lost his appetite 2-3 weeks ago with subsequent 10-15 lbs of weight loss. (General disorders) | 1 | 0
developed back problem--low back pain (given meds in ER)--chronic problem that flared up (Musculoskeletal and connective tissue disorders) | 1 | 0
More back pain the last 2 weeks. Has not seen an MD. Will see his MD this week. (Musculoskeletal and connective tissue disorders) | 1 | 0
rearranging furniture and went by the side table lamp and bumped my left leg (Injury, poisoning and procedural complications) | 1 | 0
Had a "pull" on his left hip . He thinks it was his arthritis acting up (Musculoskeletal and connective tissue disorders) | 1 | 0
Had vertigo only in the AM when stood up. (General disorders) | 1 | 0
Pt got sick with the noravirus (Infections and infestations) | 1 | 0
His Crohn's disease and LB pain was acting up. Did not see an MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
Knot on stomach. Pt had it drained @ DVAMC ER. Not sure of the actual dx. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pt came to ER @ DVAMC 2 mths ago for rib pain. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had eye surgery at the VA. (Surgical and medical procedures) | 1 | 0
Got a head cold. (Infections and infestations) | 1 | 0
Pt fell while carrying gardening tools in her yard. Landed on her left side and hurt her left knee. (Injury, poisoning and procedural complications) | 1 | 0
Went to local ER for stomach pain - diagnosed with kidney stones. (Renal and urinary disorders) | 1 | 0
Had Moh's surgery on right ear at Duke. (Surgical and medical procedures) | 1 | 0
prostate enlarged, now needs to catheterize self And "kidneys are trying to shut down" (Renal and urinary disorders) | 0 | 1
stood up too fast, didn't have anything to hold onto, lost balance and fell. No injured. (Injury, poisoning and procedural complications) | 0 | 1
Got out of bed too quickly, got dizzy, and fell on the floor--"was lucky didn't hurt anything". (Injury, poisoning and procedural complications) | 0 | 1
Several months ago, "knees gave out from under" him while going up steps. Not injured. (Musculoskeletal and connective tissue disorders) | 0 | 1
Has melanoma on back of knee on left leg--had biopsy, to have melanoma removed today. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
"Eyes are getting weaker because of medicine." Had to get new glasses in April. (Eye disorders) | 0 | 1
Underwent procedure in which they stopped his heartbeat to check function and rhythm- (Cardiac disorders) | 0 | 1
Stepped over shoe string and fell over. (Injury, poisoning and procedural complications) | 0 | 1
Corn on right foot / third toe (Skin and subcutaneous tissue disorders) | 0 | 1
Leaving a restaurant , caught foot on the curb, and fell landing on hands and knee-- abrasions. (Injury, poisoning and procedural complications) | 0 | 1
Had a stomach virus for one day. (Infections and infestations) | 1 | 0
Going into the bathroom door and slipped on something that was lying on the floor (Injury, poisoning and procedural complications) | 1 | 0
Rock bruised bottom of right foot while camping. Not sure what happened. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had a stomach sickness for 2-3 days, 3 weeks ago. Did not see an MD. (Infections and infestations) | 1 | 0
Had a cold for 7-10 days. Did not see an MD. (Infections and infestations) | 1 | 0
Infection in the right eye (Infections and infestations) | 1 | 0
Pt saw In VA ER for confusion & indigestion, & SOB. Received neb tx. Has COPD. (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Both feet swollen since two weeks ago. Saw MD at the VA (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain and swelling of left leg. Saw MD phlebitis. (Vascular disorders) | 1 | 0
Came down with a cold while on a cruise. No exercise so far. (Infections and infestations) | 1 | 0
Had an abscessed tooth pulled. (General disorders) | 1 | 0
Fell yesterday, did not see an MD. Feels lightheaded when standing up (General disorders) | 1 | 0
Been having some dizziness, on/off, when turning in bed or turning his head when standing. (General disorders) | 1 | 0
Left leg stays numb all the time and feels like "walking on rubber" - is getting worse. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had some chest pressure, 2-3x, while lying in bed. (Cardiac disorders) | 1 | 0
Had chest pressure, while shopping. (Cardiac disorders) | 1 | 0
Left leg is "giving out" more nowadays. (Musculoskeletal and connective tissue disorders) | 1 | 0
Patient seen by the Dermatology for multiple boils and increased SOB. (Skin and subcutaneous tissue disorders) | 1 | 0
Got the flu. Went to the VA ER and diagnosed with a post-viral COPD flair (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Had out-patient procedure to remove fluid from cyst on his left kidney. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Right knee OA flared up for 5 days. Got meds - doing OK now. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had second cataract removed around September. (Surgical and medical procedures) | 1 | 0
Sick with a stomach virus for 2 days. (Infections and infestations) | 1 | 0
Had cataract removed around August. (Surgical and medical procedures) | 1 | 0
Moh's surgery on the nose. (Surgical and medical procedures) | 1 | 0
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
had back spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Kidney stones . Went to the local ER in Morehead. Rx= pain medication. (Renal and urinary disorders) | 1 | 0
Stomach virus for 2-3 days. Feels OK now. (Infections and infestations) | 1 | 0
Had prostate procedure. (Surgical and medical procedures) | 1 | 0
Has had an URI for 7-10 days (Renal and urinary disorders) | 1 | 0
Pain in left leg/foot from DJD in LB (10 year problem). (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt reported to the local ER with a swollen and purple-blue little finger on right hand (General disorders) | 1 | 0
The hernia is still very bothersome. He is waiting for surgery. (Musculoskeletal and connective tissue disorders) | 1 | 0
Two Melanoma cancers removed off of back of his left shoulder. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pain in right knee - not exercise related (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt discovered fluid in both legs Received Lasix for 3 days. (Vascular disorders) | 1 | 0
Arthritis in right knee has been more painful in the last 3 months. Saw doc but not hospitalized. (Musculoskeletal and connective tissue disorders) | 0 | 1
Caught foot on 3 steps off a deck, and rolled his ankle--landed on hip and shoulder (Injury, poisoning and procedural complications) | 0 | 1
Knee pain has gotten worst. No activity started it, just chronic pain. Did not see doc. (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell 4-5 days ago when he slipped on rug at home. A little hurt on left side. (Injury, poisoning and procedural complications) | 1 | 0
Slid out of bed. A little sore in the thighs. Used crutches /cane for 2 days. (Injury, poisoning and procedural complications) | 1 | 0
Was told a couple of months ago that his prostate cancer has returned. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Patient continues to have a lot of pain in both knees and in R foot. (Musculoskeletal and connective tissue disorders) | 1 | 0
Feels sick today due to stopped using ETOH (Metabolism and nutrition disorders) | 1 | 0
OA in both knees has been flaring up. (Musculoskeletal and connective tissue disorders) | 1 | 0
Increased back pain. (Musculoskeletal and connective tissue disorders) | 1 | 0
Changes in blood pressure and pulse yesterday made him call his local MD who changed his medications (Cardiac disorders) | 1 | 0
His LBP has been acting up the last four weeks. This time on the right side. Discussed with his PCP (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell on his butt when he tripped on the rug inside the door. Caught himself on his right wrist (Injury, poisoning and procedural complications) | 1 | 0
Went to ER at the VA for cough - X-rates showed no pneumonia. Treated for allergies (Immune system disorders) | 1 | 0
Prescribed antibiotics for UR infection and to call back in 3 weeks. (Infections and infestations) | 1 | 0
His back pain has been acting up the last 3 weeks. (Musculoskeletal and connective tissue disorders) | 1 | 0
More SOB when walking outdoors for the last month. (Respiratory, thoracic and mediastinal disorders) | 1 | 0
The osteoarthritis and wear on his knee has been getting gradually, but significantly worse (Musculoskeletal and connective tissue disorders) | 0 | 1
Fell/slipped on water in the grocery store and hurt right hip and arm. had X-rays done on hip (Injury, poisoning and procedural complications) | 1 | 0
To the ER decreased energy and SOB with pain to both legs. Released due to no clinical findings. (General disorders) | 1 | 0
very bad cold, went to ED (Infections and infestations) | 1 | 0
diagnosed with right leg blockage from the ankle up to the stomach. Has a vascular app. (Vascular disorders) | 1 | 0
Still hurts "all over" (the body), more so past month, especially knees and hips. (Musculoskeletal and connective tissue disorders) | 1 | 0
Got a cramp in both calves while doing toe raises. Just one episode. (Musculoskeletal and connective tissue disorders) | 1 | 0
Experiencing more pain in the left hip now. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in legs is worse. (Musculoskeletal and connective tissue disorders) | 1 | 0
On 8/9 he had out pt procedure to remove scar tissue in knee that built up after his knee surgery (Musculoskeletal and connective tissue disorders) | 0 | 1
Twisted her right knee on when she grabbed the storm and landed on the step. (Injury, poisoning and procedural complications) | 1 | 0
The severe muscle pain in the legs and arms/shoulders lasted until 3-4 days ago. Did not see the MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
hip isn't doing as well" clarified as "arthritis", "can't walk as well, hurts worse" (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, in thigh muscles and behind the knees, (R worse), since 2 weeks. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had a bad cold for almost a week. No MD visit. (Infections and infestations) | 1 | 0
While at VA he got dizzy, fell, was not injured, told he was dehydrated. (General disorders) | 1 | 0
Getting dizzy more often nowadays and eyes are blurry on/off. Is seeing his Eye MD regularly. (Eye disorders) | 1 | 0
Felt dizzy and had a presyncopal episode in front of the pharmacy at the VA. (General disorders) | 1 | 0
Had a cold with fever last week. Got stomach pain/vomited - feels better now. (Infections and infestations) | 1 | 0
About a week ago, had a drain put in his eye to reduce pressure due to glaucoma. (Eye disorders) | 1 | 0
More pain in joints and muscles since last call. Has not seen his MD yet (Musculoskeletal and connective tissue disorders) | 1 | 0
While repairing a fence, got dizzy and just fell. Not injured. (Injury, poisoning and procedural complications) | 1 | 0
Walking out in yard, turned, got dizzy, and fell. Not injured. (Injury, poisoning and procedural complications) | 1 | 0
Feels he is getting weaker - more OA pain in legs. (Musculoskeletal and connective tissue disorders) | 1 | 0
Diagnosed with sleep apnea a couple of weeks ago by his local MD. Received a C-pap 3 days ago. (General disorders) | 1 | 0
Degenerative arthritis. Has "deteriorate d gradually over the last couple of years". (Musculoskeletal and connective tissue disorders) | 1 | 0
Had a cold for two weeks. No MD visit. (Infections and infestations) | 1 | 0
Kidney stones. (Renal and urinary disorders) | 1 | 0
Fell on the backdoor steps (ice). Bruises "all over" but otherwise OK. (Injury, poisoning and procedural complications) | 1 | 0
Belly aches. (Gastrointestinal disorders) | 1 | 0
Slipped on pine straw- no injury- got back up and finished playing golf. 8 mos ago (Injury, poisoning and procedural complications) | 0 | 1
emergency app for a perirectal growth. He was referred to surgery for drainage. Discharged to home. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aggravated an old back injury- lifting building materials at work. (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain for a month after bending over at work - construction work. to a chiropractor. (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell in the post office parking lot when his left knee gave out stepping off the curb (Injury, poisoning and procedural complications) | 1 | 0
Injured the right side of his rib cage while lifting something heavy at work. (Injury, poisoning and procedural complications) | 1 | 0
Diagnosed with sleep apnea. (General disorders) | 1 | 0
weight gain r/t medicine. He has been on this medicine for years, take this medicine when I get sick (Metabolism and nutrition disorders) | 1 | 0
Upper respiratory infection. Very SOB. No exercises. (Infections and infestations) | 1 | 0
Has had a viral infection. Rx from MD. (Infections and infestations) | 1 | 0
Fosamax medication flared up arthritis. (Musculoskeletal and connective tissue disorders) | 0 | 1
Was at the beach and was walking back to the hotel. Stepped on thick sand lost my balance and fell (Injury, poisoning and procedural complications) | 1 | 0
Pt has had left hip pain since the last week - says it might be his OA. (Musculoskeletal and connective tissue disorders) | 1 | 0
Legs got weaker and I stagger more. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had walking pneumonia beginning of Oct. 09. Saw doc but was not hospitalized. (Infections and infestations) | 1 | 0
Gout came back for a week. Got more medication. Feels better. (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell 4 ft off a ladder while trimming a tree. A little sore but OK. (Injury, poisoning and procedural complications) | 1 | 0
While cutting a limb off a tree, he fell from a ladder. (3M ago) (Injury, poisoning and procedural complications) | 1 | 0
Gout in big toe on R foot . Saw PCP & got meds. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had a bad cold for 2 weeks. (Infections and infestations) | 1 | 0
Was outside walking. Stepped down and fell over to the left side due to the ground being unleveled (Injury, poisoning and procedural complications) | 0 | 1
The pain in his LB has gradually moved up the spine. He has a PCP app at the VA (Musculoskeletal and connective tissue disorders) | 1 | 0
His LB pain has been acting up during the last month. Will see his PCP (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt has had more soreness in his LB the last month. He had LB surgery in 2006. (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell while biking, landed on his right hand. Went to VA ER. X-ray = 5th metacarpal fracture. (Injury, poisoning and procedural complications) | 1 | 0
Went to VA ER for a perianal abscess. General surgery lanced the abscess. (Surgical and medical procedures) | 1 | 0
Has had a stomach virus for 2 days - the whole family is sick. Has not seen an MD. (Infections and infestations) | 1 | 0
Turned his riding lawn mower over and ended up underneath. Sore all over but OK. (Injury, poisoning and procedural complications) | 1 | 0
2 "seizures" probably related to increase in dosage of medicine (Nervous system disorders) | 1 | 0
Hurt his left knee 2 weeks ago while helping his sister to move. No trauma. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Developed persistent, dry cough. No chest x-ray ordered. Pt given meds & sent home. (Infections and infestations) | 1 | 0
Got a cold. (Infections and infestations) | 1 | 0
Fell while carrying hay off a tractor and twisted his R ankle. Did not see MD. (Injury, poisoning and procedural complications) | 1 | 0
Fell off a tractor, (missed a step), 8 weeks ago and hurt/twisted his right knee. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
I was working on a tractor and bent over and picked up a front axle from the tractor (Musculoskeletal and connective tissue disorders) | 1 | 0
Was climbing a ladder, sliiped and tore rotator cuff in left shoulder. (Injury, poisoning and procedural complications) | 0 | 1
An incident of suspected gout in his foot kept him off his feet for about a week. (Musculoskeletal and connective tissue disorders) | 0 | 1
Developed "stomach/chest burning" while deer hunting. Diagnose: dyspepsia. Rx: meds. (Gastrointestinal disorders) | 1 | 0
Developed left hip pain 3 weeks ago, no trauma (thinks it is OA), lasted 2 1/2 weeks. (Musculoskeletal and connective tissue disorders) | 1 | 0
More pain in right knee and a painful corn on left foot (hard to walk). (Musculoskeletal and connective tissue disorders) | 1 | 0
Was driving a steel post and the axe hit the top of his right hand and peeled the skin off (Injury, poisoning and procedural complications) | 1 | 0
Fell off bike while riding 17 miles . Hurt his left side. Saw MD - no treatment (Injury, poisoning and procedural complications) | 1 | 0
Saw his PCP . X-ray on left heel and consult for cortisone injection (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt states at Christmas he got a cold. SOB in evenings. Saw doc, got script. (Infections and infestations) | 0 | 1
Gradually having increased pain LB and R hip pain, pt is s/p Back surgery. (Musculoskeletal and connective tissue disorders) | 0 | 1
leg cramps at night, pt reports this started couple weeks ago (Musculoskeletal and connective tissue disorders) | 0 | 1
edema in R ankle started 2 wks ago and subsided (Musculoskeletal and connective tissue disorders) | 0 | 1
injection for pain in shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
Pt has had more pain in his left ankle and knee. Has had this problem for months (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt got pain in left foot about 2 weeks ago. No trauma (Musculoskeletal and connective tissue disorders) | 1 | 0
Had extensive Moh's surgery on his nose at Duke. (Surgical and medical procedures) | 1 | 0
Twisted her left knee in the garden. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Has developed significant left knee pain. Exercise makes it worse. Arthritis has been confirmed (Musculoskeletal and connective tissue disorders) | 1 | 0
Left knee has been bothering her more since doing a lot of squatting during gardening this summer (Musculoskeletal and connective tissue disorders) | 1 | 0
The left knee pain has gotten worse. She went to the VA ER. Rx: medication, ice/rest (Musculoskeletal and connective tissue disorders) | 1 | 0
for last 2 weeks has been hurting from ankle to knee on L leg--like kicked in shins (Musculoskeletal and connective tissue disorders) | 1 | 0
Had an A-fib episode on Did not see the MD. Comes on once every 2-3 month. OK today. (Cardiac disorders) | 1 | 0
Pt. has had gradually increasing pain in right leg from knee down to ankle since beginning of Dec (Vascular disorders) | 1 | 0
Load mower off my trailer, while getting off the mower my foot got stuck on mower and fell (Injury, poisoning and procedural complications) | 1 | 0
Basal cell carcinoma removed. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Returned home from Rehab center Fell two times while walking with the cane instead of the walker. (Injury, poisoning and procedural complications) | 1 | 0
Spilled coffee in his lap while driving and got a second degree burn. (Injury, poisoning and procedural complications) | 1 | 0
Spilled coffee in his lap and got a second degree burn. Now he has seen an MD twice (Injury, poisoning and procedural complications) | 1 | 0
Had a couple of falls after going home from rehab while trying to get used to using his cane. (Injury, poisoning and procedural complications) | 1 | 0
Trouble breathing through the nose. Had surgery for his nose 6 years ago. (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ER for problems breathing. Reoccurrence of sinus polyps. CAT Scan done at DR. office. Surgery (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Woke up with difficulty breathing - allergies! Saw PCP and received meds. Doing fine now. (Immune system disorders) | 1 | 0
Pt. had a steroid injection in the spine. MD Rx= no physical activity for a week. (Musculoskeletal and connective tissue disorders) | 1 | 0
Felt nauseated /exhausted after a work-out. started having left hip pain. (Musculoskeletal and connective tissue disorders) | 1 | 0
Slipped outdoors on wet pine bark and twisted the back. Pain in lower back since then (Injury, poisoning and procedural complications) | 1 | 0
Has had a head cold. No exercises since then. (Infections and infestations) | 1 | 0
Flare-up of his ulcer. (Gastrointestinal disorders) | 1 | 0
Going out my back door and slipped on the steps, hit my right elbow and elbow swelled up. (Injury, poisoning and procedural complications) | 1 | 0
He slipped and hit R elbow on the rail in Feb. 09, "during the last snow fall" (Injury, poisoning and procedural complications) | 1 | 0
Feels that his "weak spells" are coming on more often nowadays. (Musculoskeletal and connective tissue disorders) | 1 | 0
Gout pain . First in left, then in right ankle. (Musculoskeletal and connective tissue disorders) | 1 | 0
Very sick with upper respiratory and prostate infection for 2 weeks. (Infections and infestations) | 1 | 0
Was rear-ended. Drove himself to the ER (not VA). Was pronounced OK. (Injury, poisoning and procedural complications) | 1 | 0
Was stepping off my deck and my dog jumped down on the step I was going to. I fell (Injury, poisoning and procedural complications) | 1 | 0
Bilateral hip pain/numbness the last 2 weeks when walking/standing. From the MVA? (Musculoskeletal and connective tissue disorders) | 1 | 0
Severe headaches and back pain since the traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Still has the cold that started when he was here (Infections and infestations) | 1 | 0
More bilateral hip pain since driving long distances (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in both hips has been worse. Very hard time to sleep. (Musculoskeletal and connective tissue disorders) | 1 | 0
Sick with a virus. No exercise. (Infections and infestations) | 1 | 0
Hips are still bothering him. (Musculoskeletal and connective tissue disorders) | 1 | 0
L hip has started hurting. (Musculoskeletal and connective tissue disorders) | 1 | 0
Ache in R arm for two weeks. Sounds like a nerve pain. Has not seen his MD for it. (Musculoskeletal and connective tissue disorders) | 1 | 0
Both feet swollen up to the ankles, L more than the right. Better now (Musculoskeletal and connective tissue disorders) | 1 | 0
Tingling down right arm, just above elbow. Comes and goes. (Musculoskeletal and connective tissue disorders) | 1 | 0
In the hospital for 4 days due to mental health reasons. (Psychiatric disorders) | 1 | 0
Had the flu the last 2 weeks. (Infections and infestations) | 1 | 0
Fell on ice and hit back of head (Injury, poisoning and procedural complications) | 0 | 1
Flu virus, bronchitis and pneumonia. Also had fluid in R inner ear. (Infections and infestations) | 0 | 1
Stomach virus. (Infections and infestations) | 1 | 0
Was going outside to get dog food and tripped over the end of the weed eater. (Injury, poisoning and procedural complications) | 0 | 1
When I bend over a little bit I feel pain in my lower back (Musculoskeletal and connective tissue disorders) | 0 | 1
Stiffness in right shoulder on/off for the last six month due to lifting heavy bags at work. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had some discomfort in his left hip and knee for a while - comes and goes. (Musculoskeletal and connective tissue disorders) | 1 | 0
he fell on hand when trying to catch himself. Hurt R thumb. Did see a doctor. (Injury, poisoning and procedural complications) | 1 | 0
Mid April- at gym pulled tendon in shoulder/rotator cuff. (Musculoskeletal and connective tissue disorders) | 1 | 0
His kidneys have been failing the last several month, worse now the last two month. (Renal and urinary disorders) | 1 | 0
Pulled a muscle in his right thigh/hip two days ago while adjusting a rug at home. (Injury, poisoning and procedural complications) | 1 | 0
Pain from right sciatic nerve . The diagnosis: Spinal stenosis. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has a sinus infection. Taking antibiotics. (Infections and infestations) | 1 | 0
Stomach virus (Infections and infestations) | 1 | 0
gradually had more weakness on right side from waist down, has chronic LBP on/off. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt had left eye surgery at Duke clinic in Raleigh. Follow up appt. scheduled in 2 weeks. (Surgical and medical procedures) | 1 | 0
Has had a cold for 3 weeks. Saw his local MD 10 days ago and received meds. (Infections and infestations) | 1 | 0
Have had vision problems with his left eye for several months. Has seen many eye MDs. (Eye disorders) | 1 | 0
For the last 4-5 weeks, his right hip has been bothering him when walking. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt. has chronic LBP on/off. (Musculoskeletal and connective tissue disorders) | 1 | 0
When answering phone, tripped over feet. Fell to the floor but wasn't injured. (Injury, poisoning and procedural complications) | 0 | 1
Problems with arms from nerve pain (ongoing) started UNK. (Nervous system disorders) | 0 | 1
Had skin cancer removed from his back at the VA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
cold (Infections and infestations) | 0 | 1
Fell at work 3 weeks ago. Hurt right hand and wrist. Saw a local MD x 2. Received a splint. (Injury, poisoning and procedural complications) | 1 | 0
While exercising, tripped jumping up some stairs and injured his pinky finger. There is no break (Injury, poisoning and procedural complications) | 1 | 0
Pt presented to the VA ER with UTI/prostatitis. Received meds. Doing fine now. (Renal and urinary disorders) | 1 | 0
Has had LBP the last 2-3 weeks. Has had it before but not as painful as now (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain while playing with grandkids, saw private cardiologist 5 days later (Cardiac disorders) | 0 | 1
Oct 09 had prostate biopsy. Diagnosed with cancer. Private urologist. Cary, NC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
(Nov 09) at gym, started feeling light headed, sat on bench and slumped over. (General disorders) | 0 | 1
Woke up with LBP. Has had before. (Musculoskeletal and connective tissue disorders) | 1 | 0
hip is bothering her. Beginning about 1 1/2 months ago. Sometimes quite painful. (Musculoskeletal and connective tissue disorders) | 0 | 1
Pt passed out and hurt his left big toe. Diagnose: Gout? Rx: Scheduled for an Echo, ETT (Musculoskeletal and connective tissue disorders) | 1 | 0
Had some LBP after raking leaves and fatigue feeling like having a cold. (Musculoskeletal and connective tissue disorders) | 1 | 0
Got a bad cold. Did not see an MD. Feeling better now. (Infections and infestations) | 1 | 0
Raking leaves and strained my back. (Injury, poisoning and procedural complications) | 1 | 0
Had gout out brake for 5-6 hrs. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had the flu. (Infections and infestations) | 1 | 0
Still has severe back and neck pain. Orthopedic MD has done MRI's - shows "bone on bone". (Musculoskeletal and connective tissue disorders) | 1 | 0
His back pain has been acting up and getting gradually worse the last 3 weeks. (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilateral eye surgery (cataracts). (Surgical and medical procedures) | 1 | 0
Still has LBP with some numbness in legs. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had left eye lid surgery. (Surgical and medical procedures) | 1 | 0
Fell down the steps at church. Injured hand and leg a little bit, but did not break anything. (Injury, poisoning and procedural complications) | 1 | 0
Pt. fell on the grass 10 days ago while in the yard. Jammed his finger getting up. Is fine. (Injury, poisoning and procedural complications) | 1 | 0
Diagnosed with chronic kidney disease a week ago by local PCP. (Renal and urinary disorders) | 1 | 0
Had a bad cold for a week during Christmas. (Infections and infestations) | 1 | 0
OA pain in right knee. (Musculoskeletal and connective tissue disorders) | 1 | 0
Back condition (not new) but nervous condition in stomach. MD letter stating r/t back and spine. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has been getting cramps in lower legs the last two months. The cramps lasts for several, (2-4) days (Musculoskeletal and connective tissue disorders) | 1 | 0
Went to the ER at the VA for LBP flare which might have been triggered by moving some boxes (Injury, poisoning and procedural complications) | 1 | 0
Pt has had left knee pain the last 2 weeks thinks it came from pushing hard on the clutch (Injury, poisoning and procedural complications) | 1 | 0
Pt has had the flu for 7-8 days. Saw his local MD - no meds. (Infections and infestations) | 1 | 0
Had right eye cataract surgery. (Surgical and medical procedures) | 1 | 0
Two weeks ago his head was hyper-extended for a prolonged time which caused severe dizziness (Musculoskeletal and connective tissue disorders) | 1 | 0
Had one cataract removed in November at Rex Hospital. (Surgical and medical procedures) | 1 | 0
Pinched nerve in upper right shoulder; had to have some physical therapy for it. (General disorders) | 0 | 1
Pt's face broke out red a week ago. Doesn't know why. (Skin and subcutaneous tissue disorders) | 1 | 0
Pt woke up with acute left lower back pain radiating down the left leg. Went to the VA ER (Musculoskeletal and connective tissue disorders) | 1 | 0
Had a bad cold 10 days ago. Not seen a MD. (Infections and infestations) | 1 | 0
Pt has had headaches the last month Rx; Head CT, lab work, Naproxen. (Nervous system disorders) | 1 | 0
More pain in both shoulders and LB the last 2-3 weeks - this comes and goes. Has not seen an MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
Developed pain in the three small toes on the left foot a week ago. No injury. (Musculoskeletal and connective tissue disorders) | 1 | 0
Bad headaches and more LBP during the last few weeks (Musculoskeletal and connective tissue disorders) | 1 | 0
Last month started taking Thyroid medication. (Metabolism and nutrition disorders) | 1 | 0
Feet are worse (pain in bones) no cause. (Musculoskeletal and connective tissue disorders) | 1 | 0
Got cortisone shot from his local orthopedic for his right knee about two weeks ago (Musculoskeletal and connective tissue disorders) | 1 | 0
Right knee swollen and painful since. Saw his local MD . Had X-rays. (Musculoskeletal and connective tissue disorders) | 1 | 0
Right ankle has been bothering him on and off for a couple of weeks. Did not see an MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
R elbow pain. "Hurts at the joint" it's getting worse when he moves it. (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell in a restaurant parking lot and hurt his right wrist. Did not see an MD (Injury, poisoning and procedural complications) | 1 | 0
Abscessed tooth- pulled about 3 weeks ago. Saw a periodontist. (General disorders) | 1 | 0
Pt has a bad head cold. Has not seen an MD. (Infections and infestations) | 1 | 0
started taking niacin and has since noticed some problems with his memory being "kind of slow". (General disorders) | 1 | 0
His nose bleeding got worse last three weeks. Has had it on/off for several years (Vascular disorders) | 1 | 0
Had a couple of teeth removed (General disorders) | 1 | 0
Both heels have been given me pain. (Musculoskeletal and connective tissue disorders) | 0 | 1
He had a 48 hr "Rhino" virus last week. Did not see an MD. (Infections and infestations) | 1 | 0
stepped off curb wrong and fell onto car, got 4 stitches in nose, and 2 compression fractures (Injury, poisoning and procedural complications) | 0 | 1
Tripped and fell over a block in the dark on the farm (Injury, poisoning and procedural complications) | 1 | 0
His OA in left knee has been acting up due to squatting in the garden the last many weeks. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt sick with Pneumonia Saw his local MD. Rx: nothing except rest. Doing fine now. (Infections and infestations) | 1 | 0
"Pulled" his right shoulder three weeks ago while lifting/pulling a heavy bag at the airport (Injury, poisoning and procedural complications) | 1 | 0
On the escalator in the airport luggage got stuck and slipped at the bottom and cut right thumb. (Injury, poisoning and procedural complications) | 1 | 0
Bottom "butt" was sore due to strengthening exercise from Enhanced Fitness counselor. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has a bad cold/flu since. (Infections and infestations) | 1 | 0
Twisted his right knee when leaving the VA after an app. Discussed icing. (Injury, poisoning and procedural complications) | 1 | 0
Putting gas into my car and trip over the gas hose and fell on my knees (Injury, poisoning and procedural complications) | 0 | 1
Pt has had severe LBP for the last 3 weeks. (MVA (Musculoskeletal and connective tissue disorders) | 1 | 0
Went to due to a very bad cold with breathing problems. Diagnose: acute sinusitis. Rx: antibiotics. (Infections and infestations) | 1 | 0
Pt has had numbness and pain on his right side, from the waist all the way down to the knee (Musculoskeletal and connective tissue disorders) | 1 | 0
4 to 5 months ago started having intermittent sciatica. Just started one day- no cause. (Nervous system disorders) | 1 | 0
Pt has had gout the last five days. He has it now and then and has medication for it (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt vent to the VA ER for an URI. RX: meds. (Renal and urinary disorders) | 1 | 0
Has had some dizziness. (General disorders) | 1 | 0
Had a severe cold. (Infections and infestations) | 1 | 0
Pt had cataract surgery in right eye (Surgical and medical procedures) | 1 | 0
Pain in the joints of my thumbs. (Musculoskeletal and connective tissue disorders) | 0 | 1
The weakness from thyroid medication being stopped by local PCP. It has been restarted again. (General disorders) | 1 | 0
Pt tore his right rotator cuff again one month ago and is schedule for repeat surgery (Musculoskeletal and connective tissue disorders) | 1 | 0
OA pain in both knees the last 3 weeks - does flare up during cold weather. Did not see an MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
Hurt his right shoulder using too much weight on an upper body weight machine a month ago. (Musculoskeletal and connective tissue disorders) | 1 | 0
Saw private Dr 2 wks ago for bld work and bld in urine. enlarged prostate (Renal and urinary disorders) | 0 | 1
Had an allergic reaction after eating. Saw dermatologist at the VA again who changed meds. (Immune system disorders) | 1 | 0
Developed side effects from a change in medication (General disorders) | 1 | 0
Fell . Was working in his yard and stepped in a stump hole. He twisted left knee and fell (Injury, poisoning and procedural complications) | 1 | 0
Diagnosed with cataract in both eyes. (Eye disorders) | 1 | 0
Sick for a week with a cold. Did not see an MD. (Infections and infestations) | 1 | 0
Pt. has been sick - his whole body is sore and aching. (General disorders) | 1 | 0
Left knee pain Did a lot of yard work (Musculoskeletal and connective tissue disorders) | 1 | 0
His neuropathy has been worse the last week. Has not been walking. (Nervous system disorders) | 1 | 0
LBP. Has had it on/off for two years. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt scheduled to have right TKA at Duke a.s.a.p. Is not allowed any walking for exercise (Musculoskeletal and connective tissue disorders) | 1 | 0
Developed stingers in both feet. (Musculoskeletal and connective tissue disorders) | 1 | 0
Received results from an MRI done (before enrolling in study). Two bulging discs (L3-L5). (Musculoskeletal and connective tissue disorders) | 1 | 0
Injured left knee doing leg press at fitness club where he lives (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis in neck shoulders and hip are getting worse. (Musculoskeletal and connective tissue disorders) | 0 | 1
Breathing has gotten worse (short of breathe). (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pt heard a loud pop in his right knee when walking up a step in barn. climbing stairs is painful. (Musculoskeletal and connective tissue disorders) | 1 | 0
spell with severe nausea 10 days ago. Went to his local MD : gallbladder/pancreatitis/hepatitis? (Endocrine disorders) | 1 | 0
Did a CT scan at the VA which showed two nodules on right lung. Follow-up CT in 3 month. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Has a bad cold. Saw his MD, had Chest X-ray done and Rx antibiotics (Immune system disorders) | 1 | 0
Pain in left hip/leg . Saw his PCP. (Musculoskeletal and connective tissue disorders) | 1 | 0
He has had pain in right hip/groin. No trauma (Musculoskeletal and connective tissue disorders) | 1 | 0
Had Moh's surgery a week ago. (Surgical and medical procedures) | 1 | 0
More pain from his arthritis the last weeks, partly due to the weather. (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell in a trench he couldn't see, and hurt his upper lip. (Injury, poisoning and procedural complications) | 1 | 0
Pt has had a head cold for three weeks. Not seen an MD. (Infections and infestations) | 1 | 0
His left foot/ankle pain flared up 2 days ago (Musculoskeletal and connective tissue disorders) | 1 | 0
His back is giving him a problem 09. This has happened before but not to this extent (Musculoskeletal and connective tissue disorders) | 1 | 0
Got flu like symptoms. Received meds. (Infections and infestations) | 1 | 0
Had bilateral conjunctivitis and saw MD. Received meds. (Infections and infestations) | 1 | 0
Had a back spasm. Went to Dr. and got physical therapy. (Musculoskeletal and connective tissue disorders) | 1 | 0
L arthroscopic surgery for torn cartilage. (Surgical and medical procedures) | 0 | 1
Pt went to the VA ER for abdominal bloating, GI app. (Gastrointestinal disorders) | 1 | 0
Pt has had a headache flare up for 2-3 weeks (General disorders) | 1 | 0
Has had a bad sinus infection for 3 weeks. Went to local Urgent Care on and got antibiotics (Infections and infestations) | 1 | 0
Head cold sinus (running nose and coughing. (Infections and infestations) | 1 | 0
PT fell Hit the chair with his 4th toe on the L foot. : possible break Received a soft shoe. (Injury, poisoning and procedural complications) | 1 | 0
Sick to his stomach - very stressful situation in his life right now. Boot-camp nightmares. (Psychiatric disorders) | 1 | 0
Stomach sickness for two weeks. Has had this coming/going for many years. Did not see an MD. (General disorders) | 1 | 0
Been feeling angry and having night sweats and nightmares getting worse the last 2 weeks. (Psychiatric disorders) | 1 | 0
Received cortisone injections for pain in both shoulders, both knees and LB 10 days ago (Musculoskeletal and connective tissue disorders) | 1 | 0
His right knee (OA), has been painful the last weeks too - no Treadmill walking. (Musculoskeletal and connective tissue disorders) | 1 | 0
His OA acted up 2 weeks ago due to working out in the cold. Received injections (Musculoskeletal and connective tissue disorders) | 1 | 0
His PTSD has flared up the last 2 weeks. (Psychiatric disorders) | 1 | 0
having problems w/ sore throat and a cough, dx w/ upper respiratory infection. (Infections and infestations) | 0 | 1
Had shingles about a month ago on right side of upper chest/back area. Saw doc. (Immune system disorders) | 0 | 1
Has had a severe cold for 2 weeks. (Infections and infestations) | 1 | 0
Passed blood 2 weeks ago - this happens when in physical stress. Has not seen his MD (Renal and urinary disorders) | 1 | 0
Right knee a little swollen. Happens now and then. (Musculoskeletal and connective tissue disorders) | 1 | 0
Got a head cold (Infections and infestations) | 1 | 0
Sinus infection for 2 days. (Infections and infestations) | 1 | 0
severe pain in lower back which has increased since last visit (Musculoskeletal and connective tissue disorders) | 1 | 0
He had the flu for three weeks. (Infections and infestations) | 1 | 0
Has had a cold for a few days. (Infections and infestations) | 1 | 0
Fell and hit his head on the pavement while playing basketball with his grandchild (Injury, poisoning and procedural complications) | 1 | 0
Had scheduled hernia surgery done at the VA. Doing fine. (Surgical and medical procedures) | 1 | 0
Pt's left ear started "ringing" four weeks ago and after a week he lost all his energy. (Ear and labyrinth disorders) | 1 | 0
Woke up a week ago with left foot pain and weakness - felt like the left foot was going to give out (Musculoskeletal and connective tissue disorders) | 1 | 0
Reported to the VA ERfor a rash (tick or spider bite?) on his left upper thigh, nausea (Infections and infestations) | 1 | 0
His LBP with pain down in left leg has been acting up the last 3 days. Has not seen an MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
Caught a stomach virus. Called the MD for Rx. Feeling better today. (Infections and infestations) | 1 | 0
Got bit by a spider about 3 weeks ago and had to be put on antibiotics by his doctor. (Infections and infestations) | 1 | 0
Taken off arthritis med by his PCP. He has been in a great deal of pain since then. (Musculoskeletal and connective tissue disorders) | 1 | 0
The left hip and LB pain worse last week, (OA due to old war injury). (Musculoskeletal and connective tissue disorders) | 1 | 0
His lower back pain was acting up last week. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had a cold. (Infections and infestations) | 1 | 0
LBP after making a "bad twist". Not seen an MD. (Musculoskeletal and connective tissue disorders) | 1 | 0
less sleep due to PTSD problems and sleeping meds not working as well (Psychiatric disorders) | 0 | 1
sinus and hay fever have worsened; (Infections and infestations) | 0 | 1
Partial blindness in right eye when woke up . Had surgery for retinal detachment (Eye disorders) | 1 | 0
Tripped and fell Hit his right knee - just a bruise - has not seen the MD. (Injury, poisoning and procedural complications) | 1 | 0
pt "tripped and fell at the house". Pt states he tripped on pre-existing carpet at home. (Injury, poisoning and procedural complications) | 1 | 0
chair rolled from under me and I hit the concrete floor in my garage. I jarred my left hip. (Injury, poisoning and procedural complications) | 1 | 0
loading truck with plywood the plank slipped out of my hand and fell on my L big toe (Injury, poisoning and procedural complications) | 1 | 0
Was in a car accident - hit by a car - Went to the local hospital and checked out OK. (Injury, poisoning and procedural complications) | 1 | 0
Had some "tinkling" in his both hands, on/off, . Saw MD and checked out OK. (General disorders) | 1 | 0
Pain in left shoulder. Still doing his exercises - doesn't make it worse. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt. got chest pain/GI pain after doing heavy labor. Ruled out for MI. Diagnose: gallstones. (Gastrointestinal disorders) | 1 | 0
His chronic bronchitis flared up last week. Saw his local PCP and got antibiotics. (Infections and infestations) | 1 | 0
Has had several gallbladder attacks. Has an appointment with the GI surgeon to discuss surgery. (Gastrointestinal disorders) | 1 | 0
Pt's R knee, (torn meniscus), and left shoulder (torn rotator cuff) "flared up" a week ago (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt had laparoscopic cholecystectomy at the VA. Discharged to home the next day. (Surgical and medical procedures) | 1 | 0
5 months ago had 4 stents put in at the Durham VA. (Surgical and medical procedures) | 1 | 0
Pt's R knee OA flared up. (Musculoskeletal and connective tissue disorders) | 1 | 0
Both hands became red with blisters (chemical burn?), (Skin and subcutaneous tissue disorders) | 1 | 0
Knee and ankle. (The knee was an issue before ) and the ankle pt is unsure of what going on (Musculoskeletal and connective tissue disorders) | 1 | 0
Sore throat and sinus infection for a week. Saw PCP. Rx: antibiotics. (Infections and infestations) | 1 | 0
Removed a "pre-cancerous melanoma" from the R chest area a few weeks ago. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Left foot pain since three weeks ago after wearing a new pair of shoes. (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had bronchitis. Saw his local PCP today. (Infections and infestations) | 1 | 0
Got bronchitis. Will see his local MD tomorrow. (Infections and infestations) | 1 | 0
was going down wooden steps which was wet from the rain and I slipped and fell (Injury, poisoning and procedural complications) | 1 | 0
Was doing my walking exercise and stepped in a pothole and tripped which tweaked my right knee. (Injury, poisoning and procedural complications) | 1 | 0
Pt hurt his right knee 10-14 days ago by twisting the knee when stepping in a hole (Injury, poisoning and procedural complications) | 1 | 0
Has had the flu. Has not seen an MD. (Infections and infestations) | 1 | 0
Heart is beginning to beat faster. (Cardiac disorders) | 1 | 0
Twisted his left ankle and the left knee when walking down the front steps of his house (Injury, poisoning and procedural complications) | 1 | 0
Working in his yard (his roses) and he fell--doesn't know why or how he fell. (Injury, poisoning and procedural complications) | 0 | 1
Pt had an accident at work where he broke and cut the ring finger on his right hand (Injury, poisoning and procedural complications) | 1 | 0
Moving some electrical wire rears, cut my right hand ring finger half way off. ER sewed it back on. (Injury, poisoning and procedural complications) | 1 | 0
Pt has had bilateral knee pain, left worse than right, for two weeks. Is now limping. No injury (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulled my right groin by lifting some wire at work. (Injury, poisoning and procedural complications) | 1 | 0
Pt had out-patient left carpal tunnel release surgery at the VA (Surgical and medical procedures) | 1 | 0
Pt. got hit in the forehead in the GYM by an exercise machine that was let go too quickly (Injury, poisoning and procedural complications) | 1 | 0
Had a tooth pulled. (General disorders) | 1 | 0
kidney stone. (Renal and urinary disorders) | 1 | 0
Depression."Was in a bad cycle for a month, month and a half" mother in law hospitalized. (Psychiatric disorders) | 1 | 0
Injured tubing down the Virgin River. Shoulder, neck, knees feet, bottom was bruised. (Injury, poisoning and procedural complications) | 1 | 0
Fell out of bed after a dream. Bruised his right knee. Did not see an MD for it (Injury, poisoning and procedural complications) | 1 | 0
Kidney stones (3) passed. All summer long. Passed most sever one "2 weeks ago". (Renal and urinary disorders) | 1 | 0
His PTSD has been acting up the last four weeks. Usually happens in the fall. (Psychiatric disorders) | 1 | 0
Got a stomach virus - feeling better now. Did not see an MD. (Infections and infestations) | 1 | 0
Passed a kidney stone. Did not see an MD. (Renal and urinary disorders) | 1 | 0
Has had a sinus infection for at week and a half in Nov/Dec. (Infections and infestations) | 1 | 0
Right knee pain when bending it. Thinks he bumped it during work (he repairs trucks). (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus /bronchitis infection . Saw MD - received medications. (Infections and infestations) | 1 | 0
Pain in left shoulder last 3 weeks from working overhead - no trauma (Injury, poisoning and procedural complications) | 1 | 0
Has been up to the VA in Virginia for 2 weeks for his PTSD. (Psychiatric disorders) | 1 | 0
Pt tripped over her dog and fell. Hurt her left side of chest - very painful. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Pulled a muscle in LB while doing the Squat the first time. (Musculoskeletal and connective tissue disorders) | 1 | 0
Saw his PCP at the VA and was declared having Diabetes II and received metformin. (Metabolism and nutrition disorders) | 1 | 0
Problem with right foot - heavy pain, could not walk. Went to the ER at the VA (Musculoskeletal and connective tissue disorders) | 1 | 0
In to the VA ER today, for hemorrhoidal bleeding. Doing OK now. (Skin and subcutaneous tissue disorders) | 1 | 0
Has had some discomfort in the chest - - last 3 days (not today) (Cardiac disorders) | 1 | 0
Pt fell on her sacrum on a grassy slope, while opening the door on her car. (Injury, poisoning and procedural complications) | 1 | 0
Could hardly move due to pain in hips for an hour cooking . Pain on/off for 3 days. (Musculoskeletal and connective tissue disorders) | 1 | 0
She has had terrible LBP She has OA in hips and a history of LBP. No trauma. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had a bad head-cold for 2 weeks. Did not see an MD. (Infections and infestations) | 1 | 0
Reported to the VA ER for a tick bite. (General disorders) | 1 | 0
Muscles feel weaker. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt has had symptoms of vertigo . PCP informed her that she might have had "mini-strokes". (Nervous system disorders) | 1 | 0
Pt developed pain in her spine and neck during a new exercise position in her yoga class (Musculoskeletal and connective tissue disorders) | 1 | 0
Has experienced side effects from flu/pneumonia shot the last couple of weeks. (General disorders) | 1 | 0
Her LBP was acting up for 2.5 weeks - feeling better now. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt got bronchitis two weeks ago. Rx: antibiotics. (Infections and infestations) | 1 | 0
Been having some dizziness. (General disorders) | 1 | 0
Pt experienced severe stomach cramps and a flare up of his colitis (Gastrointestinal disorders) | 1 | 0
Pt had a bad fall when stepping over a small gate (Injury, poisoning and procedural complications) | 1 | 0
stepped over a gate and and I fell over on my left knee, right hand and left side of my head. (Injury, poisoning and procedural complications) | 1 | 0
Pt got a virus with fever and joint ache, lasting for three days. No MD visit. (Infections and infestations) | 1 | 0
Had a cold for 3 weeks. (Infections and infestations) | 1 | 0
Stepped off a curb and hurt his back. Saw MD - Rx rest for a week. (Injury, poisoning and procedural complications) | 1 | 0
Allergy reaction last night (Immune system disorders) | 0 | 1
Arthroscopic right knee surgery. Released same day. (Surgical and medical procedures) | 1 | 0
Missed the last step walking down the stairs in his house and fell on his right side. (Injury, poisoning and procedural complications) | 1 | 0
More pain in Right knee. He is scheduled for arthroscopic knee surgery (Musculoskeletal and connective tissue disorders) | 1 | 0
Has had a cold for a week. Has not seen MD. (Infections and infestations) | 1 | 0
Primary Care Doc says he is now "Diabetic"; his highest A1c was 6.8, it is now back down to 6.7. (Metabolism and nutrition disorders) | 1 | 0
His left Plantar Fasciitis has been acting up. (Musculoskeletal and connective tissue disorders) | 1 | 0
Diagnosed with diabetes. (Metabolism and nutrition disorders) | 1 | 0
Had surgery on left ear drum (chronic ringing in ear). Out pt. (Surgical and medical procedures) | 0 | 1
More pain in the left ear than usually. (Ear and labyrinth disorders) | 0 | 1
Bil Rotator cuff problems No problems before pt is unsure if rotator cuff but its shoulder joint (Musculoskeletal and connective tissue disorders) | 1 | 0
LBP "something kicks in" started last few months. Not taking any meds. Did not see a doctor. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt was tired all the time and had a stress test done No ER Thinks it was related to the CPAP machine (General disorders) | 0 | 1
episode of Avib when he woke up in the morning. - Went to ER in Grandville Co (Cardiac disorders) | 0 | 1
More pain in left leg and LB. Scheduled for an MRIand will try to see his PCP then too. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in knees and back for the last month. He has a pinched nerve and arthritis in the knees. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain all the way down in left leg. Had an appointment with the pain clinic (Nervous system disorders) | 1 | 0
Feeling dizzy and was taking home BP. Was given HTN diagnosis. Was prescribed another medication . (General disorders) | 0 | 1
Bumped his head and got an OA flare in his LB and right hip (Injury, poisoning and procedural complications) | 1 | 0
He hurt his LB while pulling out the trash cart. (Injury, poisoning and procedural complications) | 1 | 0
Has had a bad cold for 3 weeks starting. Received antibiotics over the phone from the VA . (Infections and infestations) | 1 | 0
Had really bad cold that lasted a long time. Saw doc but not hospitalized. (Infections and infestations) | 1 | 0
Bad recurring cold. Saw his PCP and got antibiotics. (Infections and infestations) | 1 | 0
Has occasional problems with his PTSD--he calls them "episodes" (Psychiatric disorders) | 1 | 0
Sick for 10 days with URI coughing blood. (Infections and infestations) | 1 | 0
Pt fell 5 feet down in the chicken house 3 weeks ago. Hurt his right knee. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Crook in neck r/t sleeping habits -per pt (Musculoskeletal and connective tissue disorders) | 1 | 0
fell forward and hit my left eyebrow on my hard wood floor and got a one inch cut (Injury, poisoning and procedural complications) | 1 | 0
fell down 3 steps and landed on my bottom. Bruised hip and the back side of my thigh. (Injury, poisoning and procedural complications) | 1 | 0
Was outside when stepping up on brick steps missed a step and fell down landing on my back (Injury, poisoning and procedural complications) | 1 | 0
Tripped and hit his ribcage on a fence . Pain on right side. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Had stomach flu for three days twice the last weeks. Did not see an MD. (Infections and infestations) | 1 | 0
Stomach flu. (Infections and infestations) | 1 | 0
Diagnosed with diabetes in November. (Metabolism and nutrition disorders) | 0 | 1
Got dust in his eye hanging sheet rock, Conjunctivitis. Rx: gentamicin eye ointment. (Infections and infestations) | 1 | 0
Sinus infection after going on CPAP machine. (Infections and infestations) | 1 | 0
Went to the VA ER due to right knee being very tender (on the outside, above the knee cap (Musculoskeletal and connective tissue disorders) | 1 | 0
Diagnosed with right patellar -femoral tendonitis/patellar-femoral syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Got a sinus infection and went to the urgent care in Asheboro. Feels OK now. (Infections and infestations) | 1 | 0
Hurt his R knee (has OA), while walking on a gravel road to pick up the mail. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt went to the local ER with stomach cramps (Gastrointestinal disorders) | 1 | 0
Broke a tooth this morning. Will go back to the VA dentist (General disorders) | 1 | 0
Has had a bad sinus infection for 10 days. Not been able to use his CPAP - feeling very tired. (Infections and infestations) | 1 | 0
Sick with a cold and sinus infection. Went to local urgent care and received antibiotics. (Infections and infestations) | 1 | 0
Burned his left hand while pressure washing a week ago. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Pt reported to the VA ER for return of cough. Rx: Augmentin. (Infections and infestations) | 1 | 0
Has had cold for a week. Did not see an MD. (Infections and infestations) | 1 | 0
Begin to have hip pain. (Musculoskeletal and connective tissue disorders) | 1 | 0
Left shoulder has been bothering him the past month. OA. (Musculoskeletal and connective tissue disorders) | 1 | 0
Both ankles and feet are more swollen since his medication was changed (Musculoskeletal and connective tissue disorders) | 1 | 0
"electric shocks" going through his body. Not a new experience, on both sides of body now. (General disorders) | 1 | 0
Developed a naval hernia 3 weeks ago when lifting heavy objects (Musculoskeletal and connective tissue disorders) | 1 | 0
Presented to the VA ER for an URI. Rx medication. Scheduled for a fistulotomy (Renal and urinary disorders) | 1 | 0
Has had a cold since he got the flu shot 10 days ago. (Infections and infestations) | 1 | 0
Pt developed left sided chest pain while watching TV, Diagnose: no ischemia. (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pt bitten by a tick. Symptoms: nausea and sweats. Made an app with VA PCP. Rx: antibiotics. (Infections and infestations) | 1 | 0
Has had migraine and nausea for the last two weeks. Has medication for it. (General disorders) | 1 | 0
Pt went to the VA ER for LBP . Diagnose: muscular strain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell inside a closet at home . Injured his left shoulder. (Injury, poisoning and procedural complications) | 1 | 0
Fell trying to show grandson how to ride scooter--hit handlebars and bruised his ribs (Injury, poisoning and procedural complications) | 1 | 0
Took a tumble in bedroom and injured left shoulder--did see MD for this. (Injury, poisoning and procedural complications) | 1 | 0
Has had a head cold since last week. Has not seen MD. (Infections and infestations) | 1 | 0
Pt was diagnosed with Diabetes 3 weeks ago. (Metabolism and nutrition disorders) | 1 | 0
Has been having dizzy spells with increased vision problems and neuropathy. (Nervous system disorders) | 0 | 1
Walked into a trailer hitch- early April. Really bruised up his leg. Not exercising at time. (Injury, poisoning and procedural complications) | 0 | 1
Developed stress fracture in right foot, which cut tendons in right foot--had surgery to repair (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain is getting worse. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulled quad muscle a couple of months ago while doing chores. (Injury, poisoning and procedural complications) | 1 | 0
Pt fell when working on a bridge and hurt his right hip a little. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
Got a bad cold last week. Has not seen an MD. Feeling better now. (Infections and infestations) | 1 | 0
Pt called and said he fell off an 8 ft ladder on and broke his left heel bone. (Injury, poisoning and procedural complications) | 1 | 0
Started having pain in R arm around elbow joint in AM. Goes away during the day. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had the flu/head cold for a few days 3 weeks ago. Did not see an MD. (Infections and infestations) | 1 | 0
Pt has had bladder problems/pain for several weeks. (Renal and urinary disorders) | 1 | 0
Stomach pain , (comes and goes due to previous radiation). Did not see a MD. (Gastrointestinal disorders) | 1 | 0
Pt got "too hot and nauseated" a month ago when walking outdoors during hot weather. (Musculoskeletal and connective tissue disorders) | 1 | 0
tripped over the back ramp of truck. Fell forward of both hands and bruised them. (Injury, poisoning and procedural complications) | 0 | 1
Incontinence is worse. (Renal and urinary disorders) | 0 | 1
He has had LBP for the last four weeks after twisting the back while lifting a heavy object at work (Injury, poisoning and procedural complications) | 1 | 0
His back problem has been acting up again with left foot feeling numb (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain. Started 3 weeks ago. Not a new problem, "put me out of work for a week, (Musculoskeletal and connective tissue disorders) | 1 | 0
Injured his back--. The LBP was caused by a lift/twist movement. (Injury, poisoning and procedural complications) | 1 | 0
Tendonitis on outside left leg, has had it for a month, but it has been more painful. (Musculoskeletal and connective tissue disorders) | 1 | 0
Still having a flare of his PTSD. Has a MH app. (Psychiatric disorders) | 1 | 0
Blister on back of right heel after getting new shoes. (General disorders) | 1 | 0
Foot pain - plantar fasciitis. (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis in right elbow. (Musculoskeletal and connective tissue disorders) | 1 | 0
More pain in R hip & L knee. Went to the VA ER. Rx: Discontinue the statin medication. (Musculoskeletal and connective tissue disorders) | 1 | 0
Woke up one night a week ago with pain in both elbows -comes and goes. Has had it before (Musculoskeletal and connective tissue disorders) | 1 | 0
Stepped on a nail. No med record for Doc visit at VA (Injury, poisoning and procedural complications) | 1 | 0
Still a lot of chronic pain. (General disorders) | 1 | 0
Stomach virus for 24 hrs. (Infections and infestations) | 1 | 0
His bilateral knee pain has gotten worse during the course of the last two weeks (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee pain is more severe--will have right knee replaced this Thursday (Musculoskeletal and connective tissue disorders) | 1 | 0
Both his knees were very sore and swollen after the walk on Sunday (Musculoskeletal and connective tissue disorders) | 1 | 0
Saw Ortho and received HA injections in both knees. (Musculoskeletal and connective tissue disorders) | 1 | 0
Strained my back/ Was outside putting corn out for the deers and pulled my back. (Injury, poisoning and procedural complications) | 1 | 0
Has had cramps in arms and legs for 3 weeks - saw his local MD 2 weeks ago - received D-vitamin (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff has been bothering him more than it used to. He has to have injections regularly (Musculoskeletal and connective tissue disorders) | 1 | 0
Yesterday, banged toe really badly against a piece of furniture. Thinks he may have broken it. (Injury, poisoning and procedural complications) | 1 | 0
His allergies have been acting up the last two weeks due to the pollen season. (Immune system disorders) | 1 | 0
Went to Local MD with stomach pain. Diagnosed with hernia (Gastrointestinal disorders) | 1 | 0
Shoulder pain with cramps flared up. Saw doctor. (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemorrhoids have gotten worst- scheduled for surgery later this month. (Skin and subcutaneous tissue disorders) | 0 | 1
Stepped on hot coals with his right foot while grilling outdoors. (Injury, poisoning and procedural complications) | 1 | 0
Pt hurt his back while changing the battery in his tractor 10 days ago. went to the chiropractor. (Injury, poisoning and procedural complications) | 1 | 0
Has been very depressed for a long time. He is under the care of his MD. (Psychiatric disorders) | 1 | 0
Has had the flu for 2 weeks. Has not seen an MD. (Infections and infestations) | 1 | 0
Sick with the flu for more than a week. (Infections and infestations) | 1 | 0
Depression. (Psychiatric disorders) | 1 | 0
right foot slipped on wet grass and I fell down. The next day my back, hip and right leg was sore. (Injury, poisoning and procedural complications) | 0 | 1
Was tried to cut meat off a bone and cut left knuckle. Left hand swollen. (Injury, poisoning and procedural complications) | 0 | 1
"tingling in my fingers" started in the "last month"; cortisone shot L shoulder (pt plays tennis) (Musculoskeletal and connective tissue disorders) | 1 | 0
severe cough and left side chest pain/soreness. Diagnosed with bronchitis - Rx medications. (Infections and infestations) | 1 | 0
Admitted to the VA for atypical chest pain - pain more related to PTSD/anxiety (Psychiatric disorders) | 1 | 0
Left knee swollen, has been swollen on and off for a year. Is not feeling well (Musculoskeletal and connective tissue disorders) | 1 | 0
Left ankle sore and swollen. No injury. (Musculoskeletal and connective tissue disorders) | 1 | 0
Been feeling sick - nauseous. (General disorders) | 1 | 0
Had the flu/strep throat. (Infections and infestations) | 1 | 0
Has had a touch of flu. (Infections and infestations) | 1 | 0
PTSD flare-up. (Psychiatric disorders) | 1 | 0
2 wks ago "sick for 3 weeks" "1 week in bed" "something that was going around", "no fever" (Infections and infestations) | 0 | 1
Went to sit down on a stool in the garden and as it sunk into the dirt, he fell to the ground. (Injury, poisoning and procedural complications) | 1 | 0
Due to snow on step, slipped and fell. Other than a scrape on the hand, not injured. (Injury, poisoning and procedural complications) | 1 | 0
Urinating a lot. (Renal and urinary disorders) | 0 | 1
Pt had outpatient surgery for bladder cancer (Surgical and medical procedures) | 1 | 0
Was working in the tobacco field pulled a ligament in my right foot under the ankle. (Injury, poisoning and procedural complications) | 1 | 0
Saw local MD in July for his right foot pain went to podiatrist diagnosed with Plantar fasciitis. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pt had another UTI a month ago and saw his local MD: RX : antibiotics and referred to urologist. (Renal and urinary disorders) | 1 | 0
Developed a pain in the bottom of right heel about 2 weeks ago when walking/working all day (Musculoskeletal and connective tissue disorders) | 1 | 0
Went to the local MD for an UTI and was treated with antibiotics. (Renal and urinary disorders) | 1 | 0
He had an UTI 2 weeks ago and saw his local MD. Rx: antibiotics. (Renal and urinary disorders) | 1 | 0
Developed LBP radiating down the right leg,while painting baseboards in the house. (Musculoskeletal and connective tissue disorders) | 1 | 0
Got LBP while twisting when lifting a box. Went to local ER - drop in clinic (Injury, poisoning and procedural complications) | 1 | 0
Pt got blisters on the ball of the right footwhen walking on the beach. (Musculoskeletal and connective tissue disorders) | 1 | 0
LBP for 3 days when bending over to pick up a key from the floor . (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue and SOB during exertion since his MI. Cardiologist to schedule a nuclear ETT (Cardiac disorders) | 1 | 0
Has chronic neck pain on/off since two years. It is now getting worse. Surgery/fusion, is planned (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulled a muscle in his right leg two weeks ago when walking around in his house. (Injury, poisoning and procedural complications) | 1 | 0
Got a very bad cold - lasted for a few days. (Infections and infestations) | 1 | 0
Pt. noticed a sore muscle in right shoulder - it also looked "different". No trauma (Musculoskeletal and connective tissue disorders) | 1 | 0
Developed a Hernia. (Musculoskeletal and connective tissue disorders) | 1 | 0
walking down the stairs at home fell 14 steps. Hurt his neck and R arm. (Injury, poisoning and procedural complications) | 1 | 0
Pt reports when getting up in the morning, head hurts and he is not balanced. (General disorders) | 1 | 0
Pt presented to the VA ER for flashbacks from the Vietnam Era incident. (Psychiatric disorders) | 1 | 0
Experienced some left knee pain the last 10 days due to adding short spurs of running (Musculoskeletal and connective tissue disorders) | 1 | 0
Fell through the ceiling while in the attic. Hurt his right leg - did not see MD. (Injury, poisoning and procedural complications) | 1 | 0
Stubbed his R foot on a table one week ago, bruised his little toe. Did not see an MD. (Injury, poisoning and procedural complications) | 1 | 0
L knee bothering him "a lot more". Got knee injections again 3 total; 1 wk apart (Musculoskeletal and connective tissue disorders) | 1 | 0
Left elbow has developed a growth. Will se PCP tomorrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
More stress at work the last 3-4 weeks - "closing the books" for the year. (General disorders) | 1 | 0
The OA in his left knee and right foot has been bothering him more. (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in left hip/leg since 3 weeks ago (old injury from Vietnam) (Musculoskeletal and connective tissue disorders) | 1 | 0
Touch of flu. (Infections and infestations) | 1 | 0
Pt went to the VA ER on for his sore throat. Diagnose: mild pharyngitis. (Infections and infestations) | 1 | 0
His little toe on L foot has been painful and inflamed for 2 weeks. thinks it is an ingrown toe nail (Musculoskeletal and connective tissue disorders) | 1 | 0
Problems with L foot pain in 4th metatarsal. He reports he could not walk like he wants to. (Musculoskeletal and connective tissue disorders) | 1 | 0
Had stomach virus for a week a couple of weeks. Did not see an MD. Doing fine now. (Infections and infestations) | 1 | 0
Left knee pain down lateral side of tibia for 2 weeks. No injury. (Musculoskeletal and connective tissue disorders) | 1 | 0
His left knee has been more painful and swollen since he tried to return to work (Musculoskeletal and connective tissue disorders) | 1 | 0
Left knee still more painful and swollen. Will see a local orthopedic this week. (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No